CLINICAL TRIAL: NCT01383759
Title: Pilot Study of Bortezomib/Dexamethasone (BD), Followed By Autologous Stem Cell Transplantation and Maintenance Bortezomib/Dexamethasone For the Initial Treatment of Monoclonal Immunoglobulin Deposition Disease (MIDD) Associated With Multiple Myeloma and AL Amyloidosis
Brief Title: Bortezomib/Dexamethasone (BD), Followed By Autologous Stem Cell Transplantation and Maintenance Bortezomib/Dexamethasone For the Initial Treatment of Monoclonal Immunoglobulin Deposition Disease (MIDD) Associated With Multiple Myeloma and AL Amyloidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-061
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2019-04

CONDITIONS: Light Chain Deposition Disease (LCDD or MIDD); Light Chain and Heavy Chain Deposition Disease (LHCDD or MIDD); Monoclonal Immunoglobulin Deposition Disease (MIDD); Amyloidosis
Keywords: BORTEZOMIB (VELCADE); CYCLOPHOSPHAMIDE (CYTOXAN); DEXAMETHASONE; MELPHALAN; 11-061
MeSH Terms: conditions — Noninsulin-dependent diabetes mellitus with deafness; Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — Bortezomib; Dexamethasone

ARMS (1):
- Bortezomib/Dexamethasone (BD) , STC & Maintenance BD (Experimental): This is a pilot study to gain information and estimate the toxicity/tolerability of 1-3 cycles of BD, followed by HDM/ASCT, and maintenance therapy with BD in patients with MIDD associated with multiple myeloma and AL amyloidosis.
  Interventions: Drug: Bortezomib/Dexamethasone (BD), Followed By Autologous STC & Maintenance Bortezomib/Dexamethasone

INTERVENTIONS:
Drug: Bortezomib/Dexamethasone (BD), Followed By Autologous STC & Maintenance Bortezomib/Dexamethasone — The treatment has three phases:
  1) Initial treatment phase: This phase consists of 1-3 21-day-cycles of a combination regimen that includes bortezomib 1.3 mg/m2, IV or Subcutaneous Injection (SQ), on days 1, 4, 8, and 11; and dexamethasone 40 mg PO or IV, on days 1, 4, 8, and 11. Stem cell mobilization and HDM/ASCT. Post-ASCT consolidation/maintenance treatment phase: This phase consists of six cycles of bortezomib 1.3 mg/m2, IV or (SQ) with dexamethasone 20 mg PO or IV administered on days 1, 8, 15, and 22 every 12 weeks +/- 2 weeks. Long Term Follow Up will cease when all patients on study have fulfilled the requirements for at least five follow up appointments.

SUMMARY:
The goal of this clinical trial is to determine the toxicity and also the efficacy of a treatment that includes the following treatment: Two medications, bortezomib and dexamethasone (or BD), followed by autologous stem cell transplantation, and a prolonged course of treatment with bortezomib and dexamethasone after transplantation. This type of treatment has been very effective in multiple myeloma. However, there is little experience with this treatment in patients who have Monoclonal Immunoglobulin Deposition Disease (MIDD) or amyloidosis. The investigators and others have treated patients who have MIDD and amyloidosis with bortezomib and autologous stem cell transplantation and have had success with this treatment. But the combination of autologous transplant with BD given before and after the transplant is a new way of treating these diseases, which the investigators believe will be very effective.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = to 18
* New diagnosis of MIDD or AL amyloidosis based on pathologic findings confirmed at Memorial Sloan Kettering Cancer Center.
* Patients must show the ability to understand the investigational nature of the treatment and to give voluntary informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agree to completely abstain from heterosexual intercourse.
* Male subjects, even if surgically sterilized (i.e., status post-vasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
* Adequate organ function defined as follows: Absolute granulocytes > 1,000/mm3 and platelets > 70,000/mm3, unless low granulocyte and platelets counts are due to multiple myeloma; total bilirubin < 1.5 ULN; AST, ALT, and alkaline phosphatase < 3 times upper limit of laboratory normal; LVEF > 50% by MUGA or ECHO (the method used at baseline must be used for later monitoring); DLCO > 50 % confirmed at MSKCC; elevated creatinine is not a contraindication to enrollment
* Performance status (ECOG) < or = to 2

Exclusion Criteria:

* Patient has received other investigational drugs with 14 days before enrollment
* Prior initial treatment chemotherapy for MIDD, AL amyloidosis or multiple myeloma with the exception of one cycle of high dose dexamethasone
* Prior bortezomib treatment
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association Class III or IV heart failure (see Appendix 20.2), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Pregnant or lactating women are ineligible. A pregnancy test will be performed on each fertile premenopausal female 2 weeks prior to entry into the study. Treatment may not begin until the results of the pregnancy test are ascertained. All patients (men and women) must agree to use medically approved contraceptive measures for at least 4 weeks before starting therapy, during therapy, and for at least 3 months after therapy has stopped.
* Pre existing neuropathy, sensory or neuropathic pain findings, grade 2 or higher on the NCI CTC neurotoxicity scale.
* Concurrent active malignancy other than non melanoma skin cancers or carcinoma in situ of the cervix. Patients with previous malignancies, but which have not required anti tumor treatment within the preceding 24 months will be allowed to enter the trial. Patients with a history of a T1a or b prostate cancer (detected incidentally at TURP and comprising less than 5% of resected tissue) may participate if the PSA has remained within normal limits since TURP.
* Patients with known HIV positivity or AIDS related illness. This is based upon the possibility of increasing HIV viral load with therapy
* Any other medical condition or reason that, in the principal investigator's opinion, makes the patient unsuitable to participate in a clinical trial
* Patients with a history of hypersensitivity reactions attributed to bortezomib, boron, or mannitol.
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06-24 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hani Hassoun, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Amyloidosis: Participants with newly diagnosed AL amyloidosis
- Monoclonal Ig DepositionDisease (MIDD): Participants with newly diagnosed Monoclonal Ig DepositionDisease (MIDD)
Period: Overall Study
Arm/Group | Amyloidosis | Monoclonal Ig DepositionDisease (MIDD)
Started | 19 | 1
Completed | 19 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amyloidosis | Monoclonal Ig DepositionDisease (MIDD) | Total
Number analyzed (Participants) | 19 | 1 | 20
Age, Continuous [Median (Full Range); unit: years] | 60 [38 to 73] | 63 [63 to 63] | 60 [38 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 13 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 1 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 1 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 1 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Progression Free Survival at 12 Months
Description: of a 3-phase comprehensive treatment approach including induction with BD followed by risk adapted HDM/ASCT, followed by consolidation/maintenance therapy with BD in patients with AL amyloidosis.
Time Frame: 12 months
Population: Data were not collected for MIDD group.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Amyloidosis
Number analyzed (Participants) | 19
percentage of patients | 84 [69 to 99]

2. Primary Outcome: Participants Evaluated for Toxicity
Description: Toxicities will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Amyloidosis | Monoclonal Ig DepositionDisease (MIDD)
Number analyzed (Participants) | 19 | 1
Participants | 19 | 1

3. Secondary Outcome: To Estimate the Hematologic Response Rate
Description: [Complete Response (CR) (Normalization of the free light chain (FLC)levels and ratio; Negative serum and urine ; <5% plasma cells in bone marrow), Very Good Partial Response (VGPR) (Reduction in the dFLC (difference between involved [iFLC] and uninvolved FLC) to<4mg/dl) and Partial Response (PR)] (>/= 50% reduction in the dFLC), achieved at 12 month, and at 24 months post-initiation of treatment following the 3-phase comprehensive treatment approach.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Amyloidosis | Monoclonal Ig DepositionDisease (MIDD)
Number analyzed (Participants) | 19 | 1
Participants
  Complete Response (CR) | 7 | 0
  Partial Response (PR) | 4 | 0
  Progression of Disease (POD) | 1 | 0
  Stable Disease (SD) | 1 | 0
  Very Good Partial Response (VGPR) | 6 | 1

4. Secondary Outcome: Organ Response - Cardiac Involvement at 12 Months
Description: 12 months post-initiation of treatment following the 3 phase comprehensive treatment approach including induction with BD, followed by risk adapted HDM/ASCT, followed by consolidation/maintenance therapy with BD in patients with AL amyloidosis.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Amyloidosis
Number analyzed (Participants) | 19
Participants
  Participants without cardiac involvement | 7
  Cardiac involvement, improved | 8
  Cardiac involvement, progressed | 2
  Cardiac involvement, died during induction | 2

5. Secondary Outcome: Progression Free Survival at 24 Months
Description: following the 3-phase comprehensive treatment approach including induction with BD, followed by risk adapted HDM/ASCT, followed by consolidation/maintenance therapy with BD in patients with AL amyloidosis.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Amyloidosis
Number analyzed (Participants) | 19
percentage of patients | 68 [50 to 93]

6. Secondary Outcome: Organ Response - Cardiac Involvement at 24 Months
Description: 24 months post-initiation of treatment following the 3 phase comprehensive treatment approach including induction with BD, followed by risk adapted HDM/ASCT, followed by consolidation/maintenance therapy with BD in patients with AL amyloidosis.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Amyloidosis
Number analyzed (Participants) | 19
Participants
  Participants without cardiac involvement | 7
  Cardiac involvement, improved | 8
  Cardiac involvement, progressed | 2
  Cardiac involvement, died during induction | 2

7. Secondary Outcome: Organ Response - Renal Involvement at 12 Months
Description: as for outcome 4
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Amyloidosis
Number analyzed (Participants) | 19
Participants
  No renal involvment | 7
  Renal involvment, improved | 9
  Renal involvment, profressed | 2
  Renal involvment, died | 1

8. Secondary Outcome: Organ Response - Renal Involvement at 24 Months
Description: as for outcome 6
Time Frame: 24 months
Population: 1 participants died at the previous 12 month follow up point
Measure: Count of Participants; unit: Participants
Arm/Group | Amyloidosis
Number analyzed (Participants) | 18
Participants
  No renal involvement | 7
  Renal Involvement, improved | 9
  Normal Renal Function after Kidney Transplant | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Amyloidosis | Monoclonal Ig DepositionDisease (MIDD)
All-Cause Mortality (participants affected / at risk) | 7/19 | 0/1
Serious Adverse Events (participants affected / at risk) | 17/19 | 1/1
Other Adverse Events (participants affected / at risk) | 19/19 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amyloidosis (N=19) | Monoclonal Ig DepositionDisease (MIDD) (N=1)
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Lung infection (Infections and infestations) | 2 | 0
Sudden death NOS (General disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amyloidosis (N=19) | Monoclonal Ig DepositionDisease (MIDD) (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 7 | 0
Alanine aminotransferase increased (Investigations) | 13 | 1
Alkaline phosphatase increased (Investigations) | 17 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 16 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 7 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
CPK increased (Investigations) | 2 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 6 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Cholesterol high (Investigations) | 9 | 0
Constipation (Gastrointestinal disorders) | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Creatinine increased (Investigations) | 12 | 1
Cytokine release syndrome (Immune system disorders) | 3 | 0
Depression (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 8 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Edema limbs (General disorders) | 5 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 2 | 0
Fatigue (General disorders) | 10 | 0
Fever (General disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Hemoglobin increased (Investigations) | 3 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 13 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 6 | 0
Hypernatremia (Metabolism and nutrition disorders) | 8 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 7 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 15 | 0
Hypokalemia (Metabolism and nutrition disorders) | 13 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 1
Hyponatremia (Metabolism and nutrition disorders) | 15 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 1
Hypotension (Vascular disorders) | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INR increased (Investigations) | 11 | 1
Infections and infestations - Other, specify (Infections and infestations) | 3 | 0
Lipase increased (Investigations) | 2 | 1
Localized edema (General disorders) | 1 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 17 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Musculoskeletal & conn tissue disorder Other, spec (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 7 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 0
Neutrophil count decreased (Investigations) | 15 | 0
Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Periorbital edema (Eye disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 1
Platelet count decreased (Investigations) | 19 | 1
Presyncope (Nervous system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Serum amylase increased (Investigations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Weight gain (Investigations) | 2 | 0
Weight loss (Investigations) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 17 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT01383759/Prot_SAP_000.pdf